CLINICAL TRIAL: NCT07320664
Title: Alcohol Counter Marketing as a Breast Cancer Prevention Strategy in Young Women
Brief Title: Breast Cancer Study Tracking Risk Awareness of Alcohol Consumption and Improving Knowledge in Young Adult Women
Acronym: B-Track
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Darren Mays, Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OSU-25089; PPI-23-007 (Other Grant/Funding Number: The Breast Cancer Research Foundation)
Record Dates: First submitted 2025-12-18; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Behavior, Risk
Keywords: cancer control; cancer prevention; alcohol
MeSH Terms: conditions — Risk-Taking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-created Messages (Experimental): Participants in the intervention arm will receive the co-created intervention content about alcohol as a risk factor for breast cancer. The investigators will deliver links to the content by text messages to participants' mobile phones.
  Interventions: Behavioral: Alcohol and Breast Cancer Risk Messages
- Control (Other): Participants in the control arm will receive text only content about skin cancer risk and prevention. The investigators will deliver links to the content by text messages to participants' mobile phones.
  Interventions: Behavioral: Skin Cancer Risk Messages

INTERVENTIONS:
Behavioral: Alcohol and Breast Cancer Risk Messages — Participants will be randomized in a 1:1 ratio to the intervention or control arm. In the intervention arm, participants will receive the co-created intervention content. The investigators co-created the intervention content, including visuals and text, through focus groups with young adult women and refined the draft content based on additional feedback from focus groups, thereby ascertaining the views of young adult women. The intervention content aligns with a conceptual framework and includes messaging with the following themes: 1) Risks of breast cancer from alcohol consumption; 2) Efficacy content promoting behavior change; 3) Relevance to young adult women; 4) Mechanisms through which alcohol consumption increases breast cancer risk; 5) Exposing the alcohol industry's deceptive marketing practices; 6) Comparisons to other behavioral risk factors for cancer.
  Arms: Co-created Messages
Behavioral: Skin Cancer Risk Messages — Participants in the control arm will receive text only content about skin cancer risk and prevention. This is based on intervention trials in other cancer prevention areas (e.g., tobacco) where the investigators used this type of control, provides a contact-matched comparison relative to the intervention arm, and ensures consistency of the protocol (e.g., timing of completion and content of measures to be completed) across the trial arms.
  Arms: Control

SUMMARY:
This randomized trial aims to test the effects of co-created breast cancer counter marketing intervention messages for reducing alcohol consumption and impacting awareness and beliefs about the breast cancer risks from alcohol consumption in young adult women.

DETAILED DESCRIPTION:
This is an experimental behavioral study that builds upon prior work that engaged young adult women to collaboratively co-create counter marketing intervention content designed for digital media using open artificial intelligence, text-to-image content generation platform during real-time discussions. This study will test the refined and finalized co-created intervention content in a randomized trial by measuring alcohol consumption behavior and awareness and beliefs about the breast cancer risks from alcohol consumption. Participants will be randomized in a 1:1 ratio to the intervention arm or to a control arm. Participants in the intervention arm will receive the co-created intervention content twice a week for 6 weeks. Participants in the control arm will receive text only content about skin cancer risk and prevention for the same duration and dose. Up to 10% of participants from each trial arm will be randomly selected to wear a wrist-worm transdermal alcohol biosensor to capture an objective biochemical measure of alcohol consumption remotely.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth.
* Age 18-25 at enrollment.
* Report drinking alcohol at least once in the past 30 days.
* Not pregnant or intending to become pregnant by self-report.
* Reside in Ohio, Michigan, Illinois, Wisconsin, or New Jersey.
* Willing to complete procedures.
* Able to complete procedures a, b, or c:

  1. Can read, write, and converse in English.
  2. Has a personal mobile smartphone with texting capabilities to receive text messages that may contain text and images.
  3. For the subsample who will wear the BACTrack sensor, they must have an iPhone. At the time of this protocol, the BACTrack skyn app is only compatible with iPhones. If this expands to Android phones over the course of the study, Android phones will be eligible.

Exclusion Criteria:

* Assigned male at birth
* Ages <18 or >25 at enrollment
* Do not report drinking alcohol at least once in the past 30 days
* Pregnant or intending to become pregnant by self-report.
* Do not reside in Ohio, Michigan, Illinois, Wisconsin, or New Jersey.
* Not willing to complete procedures.
* Unable to complete procedures.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 12 weeks post intervention
  Alcohol consumption will be measured using the Timeline Follow Back, a valid self-report measure of daily alcohol consumption over the past 4 weeks. The Timeline Follow Back captures alcohol consumed each day in the past 4 weeks. The measure is administered at the end of the intervention, 4 weeks post intervention, and 12 weeks post intervention. Lower alcohol consumption is considered a better outcome.
Daily Alcohol Consumption | 12 weeks post intervention
  Daily alcohol consumption will be measured using Ecological Momentary Assessments, brief daily questions sent to participants' mobile phones that participants answer about whether they drank alcohol and, if so, how much. Daily assessment periods capture alcohol consumption from the end of the intervention to 4 weeks post-intervention, and from 8 weeks to 12 weeks post intervention. Lower daily alcohol consumption is considered a better outcome.
Intentions to Reduce Alcohol Consumption | 12 weeks post intervention
  Intentions to reduce alcohol consumption will be measured with two valid self-report items on a 1-4 scale. The items are averaged to create an overall score. Higher intentions to reduce alcohol consumption is considered a better outcome. The measure is administered at the end of the intervention, 4 weeks post intervention, and 12 weeks post intervention.
Alcohol and Breast Cancer Risk Beliefs | 12 weeks post intervention
  Alcohol and breast cancer risk beliefs will be measured using 2 valid self-report items on a 1 to 7 scale. Items will assess perceived risk of breast cancer from drinking alcohol and worry about the harm of breast cancer from drinking alcohol. The items are averaged to create an overall score. Higher risk beliefs are considered a better outcome. The measure is administered at the end of the intervention, 4 weeks post intervention, and 12 weeks post intervention.
Alcohol and Breast Cancer Efficacy Beliefs | 12 weeks post intervention
  Alcohol and breast cancer efficacy beliefs will be measured using 2 valid self-report items on a 1 to 7 scale. Items will assess confidence that reducing drinking can lower breast cancer risks and perceived reduction in breast cancer risk from reducing drinking. The items are averaged to create an overall score. Higher efficacy beliefs are considered a better outcome. The measure is administered at the end of the intervention, 4 weeks post intervention, and 12 weeks post intervention.
Awareness of the Risks of Breast Cancer from Drinking Alcohol | 12 weeks post intervention
  Awareness of the breast cancer risks from drinking alcohol will be measured using a single valid self-report item on a 1 to 5 scale. The item measures agreement or disagreement that drinking alcohol increases the risk of breast cancer. Higher values are considered better outcomes. The measure is administered at the end of the intervention, 4 weeks post intervention, and 12 weeks post intervention.
Transdermal Alcohol Concentration | 12 weeks post intervention
  Transdermal alcohol concentration will be measured with wearable biosensors in a subsample of up to 10% of participants. The biosensors capture drinking days confirmed by transdermal alcohol consumption. Fewer drinking days are considered a better outcome. Participants will wear biosensors consumption from the end of the intervention to 4 weeks post-intervention, and from 8 weeks to 12 weeks post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mays, MPH, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from self-report measures and transdermal alcohol concentration biosensors will be deposited in the Inter-university Consortium for Political and Social Research (ICPSR). ICPSR will make the research data from this project available to the broader social science research community as public-use data files. These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, may be accessed directly through the ICPSR website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The research data from this project will be supplied to ICPSR at the time of publication of the relevant results or at the end of the project period on July 1, 2027, whichever is sooner, so that any issues surrounding the usability of the data can be resolved. Data files will be permanently findable and identifiable (no end date) by assignment of a persistent unique identifier (a DOI) upon their availability in the repository. Delayed dissemination may be possible. The Delayed Dissemination Policy allows for data to be deposited but not disseminated for an agreed-upon period (typically one year).
Access Criteria: After agreeing to Terms of Use, users with an ICPSR MyData account and an authorized IP address from a member institution may download the data, and non-members may purchase the files.

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu